CLINICAL TRIAL: NCT02122978
Title: Comparing Mindfulness Based Cognitive Therapy and Mindfulness Based Self-compassion Therapy: Understanding What Works Psychologically and Physiologically in a Randomized Study in Dermatology
Brief Title: Comparing Mindfulness Based Cognitive Therapy and Mindfulness Based Self-compassion Therapy in a Psoriasis Sample
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: St Vincent's University Hospital, Ireland (Other)
Responsible Party: Principal Investigator, Dr. Paul D'Alton, Dr. Paul D'Alton, St Vincent's University Hospital, Ireland
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 19/12/12 mind derm
Record Dates: First submitted 2014-04-23; First posted 2014-04-25 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2014-04

CONDITIONS: Psoriasis
Keywords: psoriasis; dermatology; mindfulness; self-compassion
MeSH Terms: conditions — Psoriasis | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mindfulness Based Cognitive Therapy (Active Comparator): Mindfulness Based Cognitive Therapy
  Interventions: Behavioral: Mindfulness Based Cognitive Therapy
- MBSCT 8 week course (Experimental): Mindfulness Based Self Compassion Therapy
  Interventions: Behavioral: Mindfulness Based Self Compassion Therapy
- Mindfulness Based Self-Compassion - Audio guided (Active Comparator): MBSC - minimal contact
  Interventions: Behavioral: MBSC - minimal contact

INTERVENTIONS:
Behavioral: Mindfulness Based Cognitive Therapy — MBCT 8 week course delivered by trained facilitator
  Other Names: MBCT
  Arms: Mindfulness Based Cognitive Therapy
Behavioral: MBSC - minimal contact — 8 week course in Mindfulness Based Self Compassion delivered remotely by audio guided MP3
  Other Names: Mindfulness Based Self Compassion MP3
  Arms: Mindfulness Based Self-Compassion - Audio guided
Behavioral: Mindfulness Based Self Compassion Therapy — Mindfulness Based Self Compassion Therapy - 8 wee course delivered by trained facilitator
  Other Names: MBSCT
  Arms: MBSCT 8 week course

SUMMARY:
Increasing research evidence supports the effectiveness of mindfulness based interventions; however, the exact mechanisms of change are poorly understood. Some evidence proposes that self-compassion is an important mechanism of change in the effectiveness of mindfulness based interventions. The current research will evaluate and compare the effectiveness of two mindfulness meditation approaches; Mindfulness Based Cognitive Therapy (MBCT) and Mindfulness based Self-compassion Therapy (MBSCT), for individuals with psoriasis, a skin condition commonly associated with stress. Blood analyses will be conducted to assess and compare the impact of the interventions on the immune system. Self-report questionnaires will explore participants' psychological functioning (e.g. self-compassion, depression, anxiety, worry). This study will also examine whether a relationship exists between immune functioning and psychological factors. An audio-guided MBSCT programme will be piloted, with a view to trialling as a more cost-effective alternative to traditional mindfulness interventions. Findings will enable us to design more effective interventions in the future, and yield clear results regarding the existence of a definite link between immunological functioning and psychological functioning.

The main research hypothesis is that participants who complete a mindfulness based intervention will experience significantly greater psychological well-being, symptom reduction, and greater changes in telomerase and cytokine activity than individuals who only receive treatment as usual for their psoriasis.

DETAILED DESCRIPTION:
The proposed research is a randomized, multi-site, blinded comparative study of mindfulness-based cognitive therapy (MBCT), Mindfulness Based Self-compassion Therapy (MBSCT), minimal-contact MBSCT, and treatment as usual (TAU) in patients with psoriasis.

Recruitment commenced in November 2013 and continued until March 2014. Participants were recruited via the Department of Dermatology in St. Vincent's University Hospital. During weekly dermatology clinics eligible participants were identified by medical members of the Dermatology team and on expression of interest were referred to an Assistant Psychologist for recruitment purposes. In addition participants were also recruited via an advertisement placed in a national newspaper.

Eligible patients will be randomly assigned to TAU (n=25), MBCT (n=25), MBSCT (n=25), or audio-guided MBSCT (n=25).

At Time 1 (pre intervention), participants will be required to give blood (a 50ml sample, i.e., roughly 10 teaspoons), and complete self-report measures on the same day as beginning the mindfulness programme. As it has previously been indicated that cells may be sensitive to sudden changes in stress, mood and time of day (Epel, 2012), blood samples will always be taken after completing the self-report measures and at a relatively standardized time, e.g., between 3-5pm. Care will be taken to ensure that conditions are relaxed across all participants, and a 10 minute rest period between completing the questionnaires and giving blood will be enforced. Bloods can be kept at room temperate for up to 24 hours and then prepared for storage below 60 degrees Celsius until PBMC analysis is to be conducted after all samples have been collected at Time 1 (post intervention).

At Time 2, six-months and twelve-months follow-up, participants will again be required to give 50ml of blood and complete all self-report measures via an identical protocol, and analysis will be conducted again accordingly. Telomerase will be assessed using a TRAPeze EXCEL Telomerase Detection Kit. This will be complemented by flow cytometry analysis of telomere length. Serum cytokines before and after treatment will be examined by ELISA. This should give an indication of the effect of treatment on systemic inflammation. We will also examine the ability of PBMC from patients to produce proinflammatory cytokines, including IL-6, TNF, IL-1, and others associated with anxiety and depression. PBMC will be activated with innate stimulus such as LPS/zymosan. The production of cytokines will be determined by ELISA. Highly sensitive CRP is also a marker for psoriasis and will be assessed by ELISA to give an indication of overall inflammation. In regards to self-report measures, the following psychological scales will be used:

1. Hospital Anxiety and Depression Scale (HADS; Snaith & Zigmond, 1994)
2. Penn State Worry Questionnaire (PSWQ: Meyer, Miller, Metzger & Borkovec, 1990) 3 Fears of Compassion Scales (Gilbert, 2009)

4. Five Facets of Mindfulness Questionnaire (FFMQ: Baer, Smith, Hopkins, Krietemeyer & Toner, 2006) 5. World Health Organisation Quality of Life - BREF (WHO, 2004). 6. Dermatology Quality of Life Index

Addressing our research question regarding the effectiveness of the mindfulness programs involves a repeated-measures comparative group intervention design. 4x4 mixed-methods ANOVAs will be used to assess pre, post and six/twelve month follow-up differences across the four experimental conditions, with group as the independent variable and psychological experience (e.g., depression, anxiety, worry, self compassion and mindfulness) or immunological activity (e.g., PBMC telomerase and cytokines) as the dependent variables. Number of hours per week practicing mindfulness during follow-up will be entered as a covariate. Effect sizes and confidence intervals will be calculated post-hoc using G*Power in order to facilitate ease of comparison between the study findings and other future studies and the relevant field of literature. Bivariate Spearman's Correlations will be conducted to examine the relationship between psychological variables and telomerase and cytokine activity on all four testing occasions, respectively. Spearman's Correlations are chosen as a suitable non-parametric correlation analysis given reports of telomerase as non-normally distributed (e.g., Epel et al., 2010; Wolkowitz et al., 2012) and inspection of our own preliminary data.

Data will be collected on four occasions; pre and post intervention and at six and twelve months follow up.

ELIGIBILITY:
Inclusion Criteria:

* adults over 18 years
* diagnosis of mild to severe psoriasis

Exclusion Criteria:

* extraneous health issues which may influence immunological activity
* Participants deemed unsuitable for MBCT or MBSCT after a psychological assessment
* previous participation in a formal 8-week mindfulness programme (e.g., MBCT, MBSR).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2013-11; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Change in immunological markers | 14 months
  Telomerase, Cytokines, C Reactive Protein will be measured in blood at 4 time points.
Psoriasis symptom control | 14 months
  Measured by Psoriasis Area & Severity Index (PASI) and drug dose reduction (if applicable)
Psychological Well-Being | 14 months
  As measured by:
  Hospital Anxiety and Depression Scale Penn State Worry Questionnaire Fears of Compassion Scales Five Facets of Mindfulness Questionnaire
Quality of Life | 14 months
  Measured by WHO QoL index and Dermatology Life Quality Index.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Vincent's University Hospital, Dublin, Dublin, Ireland